CLINICAL TRIAL: NCT03545659
Title: Childhood Acute Lymphoblastic Leukaemia: The Effect of Follow-Up Programs for Detection of Relapse. A Nordic Population-Based Cohort Study
Brief Title: Childhood Acute Lymphoblastic Leukaemia: Follow-Up
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: ALL-Relapse
Record Dates: First submitted 2018-05-17; First posted 2018-06-04 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2020-06

CONDITIONS: Precursor Cell Lymphoblastic Leukemia-Lymphoma; Recurrence
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Mode of relapse/SMN detection — Mode of relapse/SMN detection: whether the relapse/SMN was diagnosed because of symptoms of leukaemia or diagnosed at a routine visit in the outpatient clinic.

SUMMARY:
Over the past decades, advances in treatment have led to an increasing number of children who survive cancer, resulting in a growing population of childhood cancer survivors. After end of cancer treatment on common protocols survivors are enrolled in non-harmonized follow-up programs with frequent visits and blood samples. However, the evidence for the value of these follow-up programs with respect to the effect on detecting relapse and the effects on overall survival is scarce.

The aim of the study is to give a comprehensive description of the detection mode of relapsed acute lymphoblastic leukaemia (ALL), including symptoms and blood test results. Further, we aim to evaluate if the mode of detection affects survival.

DETAILED DESCRIPTION:
Investigators have identified a cohort of children with B-precursor ALL and T-ALL enrolled in the Nordic Society of Paediatric Haematology and Oncology (NOPHO) ALL-92, ALL-2000 and ALL-2008 trials and experienced a relapse or an SMN as the first event after cessation of maintenance therapy (368 patients). From medical charts and blood test results it will be decided whether the relapse/SMN was diagnosed at a routine visit (including routine blood tests) or if the relapse was diagnosed because of symptoms at a non-scheduled visit or blood test.

As the NOPHO database probably is one of the most complete databases globally, it is an advantage to perform this study as a NOPHO study.

Results of this population based relapse study will provide an evidence-based background for planning optimal and relevant follow-up programs for children after therapy of ALL treated according to contemporary Nordic ALL protocols.

The study is important and relevant in the light of today's high ALL cure rates and a need for optimal follow-up programs after cessation of ALL treatment and possible prediction of relapse.

The timing of the project is an increased focus on the clinical relevance of routine clinical follow-up of patients treated for cancer.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with pre-B or T-cell ALL in the Nordic countries (Denmark, Sweden, Norway, Finland or Iceland)
* included in the NOPHO ALL-92, ALL-2000 or ALL-2008 trials
* treated in a Paediatric Department
* developing a relapse/SMN after cessation of maintenance therapy before 31st of December 2016

Exclusion Criteria:

* hematopoietic stem cell transplantation in first complete remission

Ages: 1 Year to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: The study population will be identified in the Nordic Society of Paediatric Haematology and Oncology ALL database.
Sampling Method: Non-Probability Sample
Enrollment: 277 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
Detection mode | Investigators will review medical charts up to three months before the diagnosis of a relapse. Relapses will be categorized to be diagnosed by either a routine visit or an extra scheduled visit.
  The proportion of relapses diagnosed at a routine visit vs. relapses diagnosed at an extra scheduled visit.

SECONDARY OUTCOMES:
Survival | Time-to-Event measures (up to 23 years from date of relapse until censoring)
  Survival, by detection mode (routine or extra visit)

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Schrøder, Professor, Study Director — Aarhus University Hospital
Locations (5):
- Department of Paediatrics and Adolescent Medicine, Aarhus University Hospital, Aarhus N, Denmark
- Department of Paediatrics and Adolescent Medicine, Turku University Hospital, Turku, Finland
- The National University Hospital of Iceland, Reykjavik, Iceland
- Department of Childhood Oncology, University Hospital Tromsø, Tromsø, Norway
- Department of Paediatric Oncology, Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No